CLINICAL TRIAL: NCT03812744
Title: Neurophysiological Effects of Whole Coffee Cherry Extract in Older Adults: An fMRI Investigation
Brief Title: Neurophysiological Effects of Whole Coffee Cherry Extract in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Jennifer L. Robinson, Ph.D., Associate Professor, Auburn University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16-391 MR 1610
Record Dates: First submitted 2018-12-14; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Memory Deficits
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Intervention Model Description: Single-site, randomized, placebo-controlled, cross-over, within-subjects design. Study sessions are no more than 72 hours apart. Visits included pre-post assessments following ingestion of either placebo or WCCE.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators, participants, and the sponsor were all blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WCCE (Experimental)
  Interventions: Drug: Whole coffee cherry extract (WCCE)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Capsule [CEBOCAP]

INTERVENTIONS:
Drug: Whole coffee cherry extract (WCCE) — 100mg WCCE
  Arms: WCCE
Drug: Placebo Oral Capsule [CEBOCAP] — Silica Oxide
  Arms: Placebo

SUMMARY:
This study was designed to characterize the changes in the brain and body associated with whole coffee cherry extract (WCCE). WCCE is a patented extract of whole coffee fruit (coffee berries) from coffea arabica. Whole coffee cherries are a source of naturally occurring nutrients. There are no known side effects or allergens associated with WCCE other than that which would be associated with a consuming typical cup of coffee.

Previous studies suggest that increases in serum concentrations of both serum total and exosomal brain-derived neurotrophic factors (BDNF) may represent one of the mechanisms responsible for improved cognitive function after acute WCCE administration. Mild cognitive impairment (MCI) is an intermediate stage between the expected cognitive decline of normal aging and the more serious decline of dementia. It can involve problems with memory, language, thinking and judgment that are greater than normal age-related changes. Furthermore, MCI is associated with reduced circulating BDNF. Due to earlier studies reporting the ability of WCCE to stimulate increases in circulating and exosomal BDNF, it has been postulated that WCCE may also acutely improve cognitive function (as measured using behavioral tasks and fMRI). The purpose of this study is to extend and elucidate the findings of previous investigations by examining the acute neurophysiological effects of WCCE using blood-oxygen level dependent (BOLD) functional magnetic resonance imaging (fMRI) and magnetic resonance spectroscopy (MRS) employing a double-blind, randomized crossover design to investigate the acute effects of a single dose of WCCE or placebo (silica oxide) on neuronal activity in older participants.

ELIGIBILITY:
Inclusion Criteria:

* Complaints of memory, verified by an informant
* 55 years of age or older

Exclusion Criteria:

* MRI contraindications
* Diagnosis of Alzheimer's Disease or suspected diagnosis at the time of visit by study personnel
* Significant cerebrovascular disease
* History of cardiovascular disease
* Current or recently prescribed medication known to interfere with peripheral and/or cerebral blood flow or vascular function

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Behavioral Measures - Change in Go/No-Go Reaction Time | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Response/reaction time for each stimuli will be recorded in ms using E-Prime. Reaction times will be calculated for correct and incorrect trials separately.
Behavioral Measures - Change in N-back Reaction Time | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Response/reaction time for each stimuli will be recorded in ms using E-Prime. Reaction times will be calculated for correct and incorrect trials separately.
Behavioral Measures - Change in Go/No-Go Accuracy | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Accuracy will be determined as the number of trials correct, and errors will be classified as errors of omission or commission.
Behavioral Measures - Change in N-back Accuracy | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Accuracy will be determined as the number of trials correct.
Change in Concentration of Neurometabolites | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Magnetic resonance spectroscopy (MRS) measurements pre/post ingestion. The following are measured: glutamate, glutamine, gamma-aminobutyric acid, N-acetylaspartate, choline, creatine, glutathione, myo-inositol, aspartate, taurine, and lactate. LCModel software performed automatic quantification of in vivo proton MR spectra by analyzing spectra as a linear combination of model spectra from sequence-specific simulations. Water-suppressed spectra were eddy current corrected and quantified using the unsuppressed water signal. Cramer-Rao lower bounds were used as a measure of fit with CRLB > 50% rejected from further analysis. Metabolite concentrations were CSF-corrected, and quantified (in ppm).
Change in Blood Levels of Brain Derived Neurotrophic Factor (BDNF) | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Serum and exosomal BDNF concentrations
Blood Oxygen Level Dependent (BOLD) Changes | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Functional magnetic resonance imaging blood-oxygen-level-dependent signal changes across tasks, and during resting state

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Robinson, Ph.D., Principal Investigator — Auburn University

IPD SHARING:
Plan to Share IPD: Undecided